CLINICAL TRIAL: NCT02913612
Title: Efficacy, Safety, and Pharmacokinetics of Timolol in Infants With Infantile Hemangioma (IH)
Brief Title: Efficacy, Safety and Pharmacokinetics of Topical Timolol in Infants With Infantile Hemangioma (IH)
Acronym: TIM01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kanecia Obie Zimmerman (Other)
Collaborators: The Emmes Company, LLC (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Kanecia Obie Zimmerman, Principal Investigator, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00068212
Record Dates: First submitted 2016-08-12; First posted 2016-09-26 (Estimated); Results first posted 2022-11-15 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Infantile Hemangioma
Keywords: Hemangioma; Infantile Hemangioma; Pharmacokinetics
MeSH Terms: conditions — Hemangioma, Capillary; Hemangioma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.25% Timolol Treatment (Experimental): Subjects assigned to this arm will be randomized to 0.25% timolol for 180 days. If during the 180 days the subject is considered a treatment failure, the subject will be unblinded. If the subject is on 0.25% timolol they will be changed to 0.5% timolol.
  Interventions: Drug: 0.25% Timolol Maleate Gel Forming Solution
- 0.5% Timolol Treatment (Experimental): Subjects assigned to this arm will be randomized to 0.5% timolol for 180 days. If during the 180 days the subject is considered a treatment failure, the subject will be unblinded. If the subject is on 0.5% timolol the treating physician will decide to either continue 0.5% timolol or withdraw the subject and begin an alternative treatment.
  Interventions: Drug: 0.5% Timolol Maleate Gel Forming Solution
- Non-Intervention Group (No Intervention): Subjects assigned to this group will not receive treatment. The subject will only be photographed on the same schedule as the intervention group.

INTERVENTIONS:
Drug: 0.25% Timolol Maleate Gel Forming Solution — 50:50 Randomized 0.25% Timolol Maleate Gel Forming Solution
  Arms: 0.25% Timolol Treatment
Drug: 0.5% Timolol Maleate Gel Forming Solution — 50:50 Randomized 0.5% Timolol Maleate Gel Forming Solution
  Arms: 0.5% Timolol Treatment

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Timolol 0.25% and 0.5% doses.

DETAILED DESCRIPTION:
Primary: Describe the efficacy of 0.25% and 0.5% topical timolol maleate Gel-forming solution (GFS) as assessed through Infantile Hemangioma (IH) changes in volume.

Secondary: Describe the safety of topical timolol maleate GFS for treatment of IH.

ELIGIBILITY:
Inclusion Criteria

1. Documented informed consent from legal guardian
2. 0-84 days postnatal age at time of first study dose or when enrolled into the non-intervention cohort.
3. Clinical diagnosis of superficial cutaneous or mucosal infantile hemangioma (must include all of the following):

   1. Superficial lesion in the dermis
   2. Thin <2 mm in thickness
   3. Small >=5 cm at its longest dimension and <=10cm2
   4. Involves skin or keratinized mucosa

Exclusion Criteria

1. History of previous treatment with any pharmacologic or laser therapy for IH
2. Ongoing therapy with an oral beta blocker or oral corticosteroid (e.g., cardiac arrhythmia, adrenal insufficiency, upper airway obstruction, tetralogy of fallot (TOF), hypertension, reactive airways disease)
3. IH that requires systemic therapy (defined by dynamic complication scale >3)
4. IH of the non-keratinized mucosa
5. Infants with more than one hemangioma that requires therapy
6. Hemodynamically significant cardiovascular disease, as determined by the investigator
7. Known allergy to beta blockers or vehicle
8. Heart rate <100 beats per minute at screening visit
9. Known prenatal or postnatal diagnosis of 2nd/3rd degree atrioventricular block
10. History of Reactive Airways Disease (RAD)
11. Any condition which would make the participant, in the opinion of the investigator unsuitable for the study.

Max Age: 84 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kanecia Zimmerman, MD, MHS, Principal Investigator — Duke Clinical Research Institute; Kristin Holland, MD, Study Chair — Medical College of Wisconsin
Locations (12):
- United States (12):
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadephia, Philadelphia, Pennsylvania
  - The University of Texas Medical School at Houston, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drolet BA, Boakye-Agyeman F, Harper B, Holland K, Lewandowski A, Stefanko N, Melloni C; Pediatric Trials Network Steering Committee (See Acknowledgments for a listing of committee members.). Systemic timolol exposure following topical application to infantile hemangiomas. J Am Acad Dermatol. 2020 Mar;82(3):733-736. doi: 10.1016/j.jaad.2019.02.029. Epub 2019 Feb 18. No abstract available. PMID 30790601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants who were eligible for the study based on inclusion and exclusion criteria but whose parents declined treatment of the hemangioma constituted the non-intervention arm of the study and served as a control group
Groups:
- Historical Controls: To obtain sufficient age-matched controls, data and clinical photographs collected as part of a similar study (EudraCT 2013-005199-17) were included in the analysis of certain outcome measures as noted in the Analysis Population Description of those measures.
Period: Overall Study
Arm/Group | 0.25% Timolol Treatment | 0.5% Timolol Treatment | Non-Intervention Group | Historical Controls
Started | 44 | 51 | 10 | 36
Completed | 32 | 33 | 7 | 36
Not Completed | 12 | 18 | 3 | 0
Not completed — Lost to Follow-up | 6 | 5 | 2 | 0
Not completed — Physician Decision | 1 | 4 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 0 | 0
Not completed — Hemangioma resolved | 1 | 0 | 0 | 0
Not completed — Local IRB decision | 1 | 0 | 0 | 0
Not completed — Study drug non-compliance | 1 | 1 | 0 | 0
Not completed — Insurance issues | 0 | 1 | 0 | 0
Not completed — Needed to treat second hemangioma | 0 | 1 | 0 | 0
Not completed — Study completion criteria not met | 0 | 1 | 0 | 0
Not completed — Ineligible | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Historical Control Group: To obtain sufficient age-matched controls, data and clinical photographs collected as part of a similar study (EudraCT 2013-005199-17) were included in the analysis of certain outcome measures as noted in the Analysis Population Description of those measures.
- Total: Total of all reporting groups
Arm/Group | 0.25% Timolol Treatment | 0.5% Timolol Treatment | Non-Intervention Group | Historical Control Group | Total
Number analyzed (Participants) | 44 | 51 | 10 | 36 | 141
Age, Continuous [Mean (Standard Deviation); unit: months] | 55.2 (17.2) | 53.6 (18.7) | 58.1 (14.4) | 47.3 (11.4) | 52.8 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 5 | 26 | 96
  Male | 12 | 18 | 5 | 10 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 0 | 0 | 17
  Not Hispanic or Latino | 36 | 41 | 10 | 0 | 87
  Unknown or Not Reported | 0 | 1 | 0 | 36 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 40 | 47 | 8 | 0 | 95
  More than one race | 3 | 4 | 2 | 0 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 36 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44 | 51 | 10 | 36 | 141

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Partial Response of Hemangioma Volume as Measured by VAS (Visual Analog Scale) Within Each Treatment Arm and Compared With Untreated Controls
Description: The VAS-volume is a 100 mm scale used to independently grade hemangioma volume. -100 indicates hemangioma has doubled in size, 0 indicates no change, and +100 indicates complete shrinkage. Partial response is defined as >20% and up to 80% reduction in volumetric size of hemangioma.
Time Frame: 180 days
Population: The Historical Control group was included with the Non-intervention group. Excludes 8 participants (four in the 0.5% dosage and four in the historical placebo controls) with out come determined to be unevaluable as they have no reported VAS scores
Measure: Count of Participants; unit: Participants
Arm/Group | 0.25% Timolol Treatment | 0.5% Timolol Treatment | Non-Intervention Group
Number analyzed (Participants) | 44 | 47 | 42
Participants | 24 | 28 | 15
Statistical Analysis 1: Comparison: 0.5% Timolol Treatment vs Non-Intervention Group; Test type: Superiority; p = 0.0205, Fisher Exact; Odds Ratio, log = 2.65, 95% CI 2-sided [1.12 to 6.26]
Statistical Analysis 2: Comparison: 0.25% Timolol Treatment vs Non-Intervention Group; Test type: Superiority; p = 0.0619, Fisher Exact; Odds Ratio, log = 2.16, 95% CI 2-sided [0.91 to 5.14]
Statistical Analysis 3: Comparison: 0.25% Timolol Treatment vs 0.5% Timolol Treatment; Test type: Superiority; p = 0.6281, Fisher Exact; Odds Ratio, log = 1.23, 95% CI 2-sided [0.53 to 2.82]

2. Secondary Outcome: Number of Participants With Partial Response in Hemangioma Color as Measured by VAS (Visual Analog Scale) Within Each Treatment Arm and Compared With Untreated Controls
Description: The VAS-color is a 100 mm scale used to independently grade hemangioma color. -100 indicates hemangioma is twice as intense, 0 indicates no change, and +100 indicates complete resolution. Partial response is defined as >30% and up to 80% reduction in color of hemangioma.
Time Frame: 180 days
Population: The Historical Control group was included with the Non-intervention group. Only participants with evaluable data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.25% Timolol Treatment | 0.5% Timolol Treatment | Non-Intervention Group
Number analyzed (Participants) | 44 | 49 | 46
Participants | 32 | 34 | 19

3. Secondary Outcome: Number of Participants With Partial Response of Hemangioma Volume as Measured by VAS (Visual Analog Scale) Within Each Treatment Arm
Description: as for outcome 1
Time Frame: 180 days
Population: Only participants with evaluable data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.25% Timolol Treatment | 0.5% Timolol Treatment
Number analyzed (Participants) | 44 | 47
Participants | 24 | 28

4. Secondary Outcome: Comparison of Partial Response of Hemangioma Color From Baseline to 180 Days, Within Each Treatment Arm
Description: Comparison of partial response of hemangioma color (partial response or greater as assessed by VAS-color) between the two treatment arms. Partial response: >30% and up to 80% reduction in color of hemangioma.
Time Frame: 180 days
Population: Only participants with evaluable data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.25% Timolol Treatment | 0.5% Timolol Treatment
Number analyzed (Participants) | 44 | 49
Participants | 32 | 34

5. Secondary Outcome: Change in Hemangioma Dynamic Complication Scale (HDCS)
Description: Absolute change in hemangioma dynamic complication scale from Day 0 to end of study within each treatment arm. The HDCS provides a 6-point severity grading system for 12 individual hemangioma-related complications (grade 0 represents absent to minimal; grade 5 = most severe). The total score ranges from 0-60.
Time Frame: baseline, day 180
Population: Only participants with evaluable data were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 0.25% Timolol Treatment | 0.5% Timolol Treatment | Non-Intervention Group
Number analyzed (Participants) | 44 | 48 | 10
score on a scale | 0 [-0.11 to 0.11] | -0.1 [-0.17 to 0.05] | 0 [0 to 0]

6. Secondary Outcome: Number of Participants Who Reach Partial Response, Assessed by Volume
Description: Assess time to partial response or greater by VAS-volume, comparing baseline to day 30, day 60, day 120 and day 180. Partial response: >20% and up to 80% reduction in volumetric size of hemangioma
Time Frame: 30 days, 60 days, 120 days, 180 days
Population: Only participants with evaluable data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.25% Timolol Treatment | 0.5% Timolol Treatment | Non-Intervention Group
Number analyzed (Participants) | 44 | 49 | 10
Participants
  30-Day Visit | 12 | 14 | 0
  60-Day Visit | 17 | 19 | 1
  120-Day Visit | 18 | 21 | 3
  180-Day Visit | 23 | 24 | 4

7. Secondary Outcome: Number of Participants Who Reach Partial Response, Assessed by Hemangioma Color
Description: Assess time to partial response or greater by VAS-color, comparing baseline to day 30, day 60, day 120 and day 180. Partial response: >30% and up to 80% reduction in color of hemangioma
Time Frame: 180 days
Population: Only participants with evaluable data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.25% Timolol Treatment | 0.5% Timolol Treatment | Non-Intervention Group
Number analyzed (Participants) | 44 | 49 | 10
Participants
  30-Day Visit | 17 | 20 | 0
  60-Day Visit | 19 | 21 | 2
  120-Day Visit | 25 | 28 | 4
  180-Day Visit | 29 | 30 | 5

8. Secondary Outcome: Change in Hemangioma Quality of Life (IH-QoL) Assessment for Infants
Description: Absolute change in IH-QoL score scale from Day 0 to end of study within each treatment arm. The IH-QoL score scale consists of 4 domains (physical symptom of patient, social functioning of patient, social and psychological functioning of caregiver, and emotional functioning of caregiver) and 29 items, with each item scored on a Likert scale : 0 = never a problem, 1 = almost never a problem, 2 = sometimes a problem, 3 = often a problem and 4 = almost always a problem). The total range is 0-116; the higher the total number indicates a worse outcome.
Time Frame: baseline, day 180
Population: Only participants with evaluable data were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Timolol Treatment | 0.5% Timolol Treatment | Non-Intervention Group
Number analyzed (Participants) | 43 | 46 | 10
score on a scale | 35.3 (8.8) | 37.4 (8.5) | 32.6 (3.3)

9. Secondary Outcome: Number of Serious Adverse Events and Adverse Events of Special Interest in Infants Treated With Topical Timolol Maleate
Description: Serious adverse events and adverse events of special interest from randomization to Day 180 in infants treated with topical timolol maleate (0.25% and 0.5%) GFS for the treatment of infantile hemangioma.
Time Frame: up to 270 days
Population: Only participants who received treatment and had evaluable data were included in this analysis
Measure: Number; unit: adverse events
Arm/Group | 0.25% Timolol Treatment | 0.5% Timolol Treatment | Non-Intervention Group
Number analyzed (Participants) | 44 | 49 | 0
adverse events
  AEs of Special Interest | 14 | 14 |
  Serious AEs | 3 | 2 |

10. Other Pre Specified Outcome: Pharmacokinetics (PK) Analysis Measuring Maximum Concentration of Timolol in Plasma Specimen
Description: The PK blood samples will be 1.0 ml each and collected between the following timeframes after application of Timolol: within 2 hours, 2-4 hours, 5-7 hours, 8-10 hours or 11-12 hours.
Time Frame: Up to 12 hours
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Pharmacokinetics (PK) Analysis Measuring Area Under the Curve of Timolol in Plasma Specimen
Description: as for outcome 10
Time Frame: Up to 12 hours
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Pharmacokinetics (PK) Analysis Measuring Volume of Distribution of Timolol in Plasma Specimen
Description: as for outcome 10
Time Frame: Up to 12 hours
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Pharmacokinetics (PK) Analysis Measuring Clearance of Timolol in Plasma Specimen
Description: as for outcome 10
Time Frame: Up to 12 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Any event excluding adverse events of special interest beginning more than 7 days after the last dose of study drug or last study procedure will not be reported. For participants in the treatment arm adverse events of special interest only will be reviewed and reported at 90 days after the last dose of study drug.
Description: 0 participants in the historical control arm were at risk for Adverse Events because they did not prospectively participate in this research study. Only data that had already been collected was used in this study.
Arm/Group | 0.25% Timolol Treatment | 0.5% Timolol Treatment | Non-Intervention Group | Historical Controls
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/51 | 0/10 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/44 | 2/51 | 0/10 | 0/0
Other Adverse Events (participants affected / at risk) | 31/44 | 28/51 | 4/10 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.25% Timolol Treatment (N=44) | 0.5% Timolol Treatment (N=51) | Non-Intervention Group (N=10) | Historical Controls (N=0)
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Respiratory syncytial virus bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.25% Timolol Treatment (N=44) | 0.5% Timolol Treatment (N=51) | Non-Intervention Group (N=10) | Historical Controls (N=0)
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 1 | 0 | 0 | NA
Plagiocephaly (Congenital, familial and genetic disorders) | 0 | 1 | 0 | NA
Amblyopia (Eye disorders) | 1 | 0 | 0 | NA
Eye discharge (Eye disorders) | 0 | 2 | 0 | NA
Diarrhoea (Gastrointestinal disorders) | 6 | 4 | 0 | NA
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | NA
Gastrooesophageal reflux disease (General disorders) | 3 | 1 | 0 | NA
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | NA
Teething (Gastrointestinal disorders) | 0 | 2 | 0 | NA
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | NA
Pyrexia (General disorders) | 6 | 6 | 0 | NA
Vaccination site pain (General disorders) | 1 | 1 | 0 | NA
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | NA
Bronchiolitis (Infections and infestations) | 2 | 1 | 0 | NA
Candida nappy rash (Infections and infestations) | 1 | 0 | 0 | NA
Conjunctivitis (Infections and infestations) | 3 | 0 | 0 | NA
Conjunctivitis bacterial (Infections and infestations) | 2 | 0 | 0 | NA
Coxsackie viral infection (Infections and infestations) | 1 | 0 | 0 | NA
Croup infectious (Infections and infestations) | 1 | 1 | 0 | NA
Ear infection (Infections and infestations) | 8 | 3 | 0 | NA
Eye infection (Infections and infestations) | 3 | 0 | 0 | NA
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0 | 0 | NA
Herpangina (Infections and infestations) | 0 | 1 | 0 | NA
Influenza (Infections and infestations) | 1 | 1 | 0 | NA
Nasopharyngitis (Infections and infestations) | 2 | 3 | 0 | NA
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | NA
Otitis media (Infections and infestations) | 2 | 0 | 1 | NA
Otitis media acute (Infections and infestations) | 0 | 2 | 0 | NA
Otitis media chronic (Infections and infestations) | 0 | 1 | 0 | NA
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 1 | 0 | NA
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | NA
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | NA
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 1 | NA
Viral rash (Infections and infestations) | 0 | 1 | 0 | NA
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA
Scar (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA
Crystal urine present (Investigations) | 1 | 0 | 0 | NA
Dairy intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA
Dizziness (Nervous system disorders) | 1 | 0 | 0 | NA
Hypotonia (Nervous system disorders) | 1 | 0 | 0 | NA
Somnolence (Nervous system disorders) | 2 | 1 | 0 | NA
Irritability (Psychiatric disorders) | 3 | 2 | 0 | NA
Mental status changes (Psychiatric disorders) | 1 | 1 | 0 | NA
Sleep disorder (Psychiatric disorders) | 2 | 2 | 0 | NA
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | NA
Cyanosis central (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | NA
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | NA
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | NA
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | NA
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA
Milia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | NA
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | NA
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | NA
Skin irritation (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | NA
Peripheral coldness (Vascular disorders) | 1 | 0 | 0 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT02913612/Prot_SAP_000.pdf